CLINICAL TRIAL: NCT01241916
Title: A Prospective Randomized Trial of Static-Progressive Versus Dynamic Splinting for Post-Traumatic Elbow Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Director of Research, Hand Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003P001441
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-05

CONDITIONS: Post-traumatic Stiff Elbows
Keywords: elbow, splint
MeSH Terms: interventions — Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Static-progressive splint (Experimental)
  Interventions: Device: Static-Progressive Splint
- Dynamic Splint (Experimental)
  Interventions: Device: Dynamic Splint

INTERVENTIONS:
Device: Static-Progressive Splint — Static progressive splinting is a well-established adjunct for restoring elbow motion. Such splints apply a static stress relaxation force to the elbow tissues, which is sequentially increased, as motion is achieved.
  Arms: Static-progressive splint
Device: Dynamic Splint — Dynamic splints are a popular alternative, and apply a constant prolonged force to the tissues as additional motion is achieved.
  Arms: Dynamic Splint

SUMMARY:
Primary Question: "When splinting is used to improve motion in post-traumatic stiff elbows, is there a significant difference in gains in motion achieved between static progressive or dynamic splint approaches?"

Secondary Question: "Is there a significant difference in patient compliance with static progressive versus dynamic splint use, and does this effect final ulnohumeral motion outcomes?"

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with post-traumatic elbow contractures in the Hand and Upper Extremity Service at Massachusetts General Hospital are eligible to for enrollment in this study regardless of sex, race or ethnicity.

Exclusion Criteria:

* Only English speaking patients will be eligible for the study since questionnaires have not been validated in other languages.

  * Vulnerable populations will not be recruited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-08; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Static-progressive Splint: Splint is worn three times per day for a 30-minute period. This splint uses stepwise increases in angle to apply force to contracted tissues that dissipates as the tissues stretch.
- Dynamic Splint: Splint is worn for approximately 6 to 8 continuous hours per day or night. This splint applies a consistent force to the tissues that is maintained as the tissues stretch.
Period: Overall Study
Arm/Group | Static-progressive Splint | Dynamic Splint
Started | 35 | 31
Completed | 28 | 21
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Static-progressive Splint | Dynamic Splint | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 30 | 64
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (13) | 45 (12) | 44 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 22 | 18 | 40
Region of Enrollment [Number; unit: participants]
  United States | 35 | 31 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Arc of Flexion and Extension
Description: Active ulnohumeral motion will be measured using a hand-held goniometer by the co-investigator not involved in the care of the patient at enrollment and 6 months after enrollment.
Time Frame: baseline and 6 months
Measure: Mean (Full Range); unit: Degrees
Arm/Group | Static-progressive Splint | Dynamic Splint
Number analyzed (Participants) | 28 | 24
Degrees | 39 [-10 to 85] | 40 [-15 to 70]

2. Secondary Outcome: Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire
Description: The DASH questionnaire measures arm-specific perceived disability. It contains 30 items and is scaled between zero and 100 with higher scores indicating worse upper-extremity function.
Time Frame: 12 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Static-progressive Splint | Dynamic Splint
Number analyzed (Participants) | 28 | 21
units on a scale | 26 [2 to 77] | 28 [3 to 76]

ADVERSE EVENTS:
Arm/Group | Static-progressive Splint | Dynamic Splint
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/31

LIMITATIONS AND CAVEATS:
Evaluation of <80% of enrolled patients at planned follow-up times; musculoskeletal injury patients are difficult to maintain in protocol. Some violations where enrollment/evaluation points were slightly outside the planned range of acceptable times.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No